CLINICAL TRIAL: NCT01903265
Title: A Phase 2b, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL Tablets Taken at Bedtime in Patients With Fibromyalgia
Brief Title: BEdtime Sublingual TNX-102 SL as Fibromyalgia Intervention Therapy (BESTFIT)
Acronym: BESTFIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F202
Record Dates: First submitted 2013-07-12; First posted 2013-07-19 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Primary Fibromyalgia
Keywords: pain; sleep
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNX-102 SL 2.8 mg (Experimental): Patients will take 1 tablet of TNX-102 SL sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL 2.8mg
- Placebo (Placebo Comparator): Patients will take 1 tablet of placebo sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNX-102 SL 2.8mg — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL 2.8 mg
Drug: Placebo — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo

SUMMARY:
TNX-102 capsules [formerly known as very low dose (VLD) cyclobenzaprine] at bedtime have shown promise as a treatment of fibromyalgia, but the drug required new formulation technology for bedtime use. The present trial was designed to assess the safety and efficacy of TNX-102 SL 2.8 mg tablets, taken daily at bedtime over 12 weeks to treat fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Fibromyalgia (ACR criteria)
* Male or female 18-65 years old
* For patients with major depressive disorders only: clinically stable, no suicidal risk and stable anti-depressent therapy
* Willing and able to withdraw specific therapies (ask PI)
* Medically acceptable form of contraception (female only)
* Signed informed consent

Exclusion Criteria:

* Arthritis, lupus and other systemic auto-immune diseases
* Regional or persistent pain that could interfere with assessment of fibromyalgia pain
* Bipolar and psychotic disorders
* Increased risk of suicide
* Significant clinical (cardiac, systemic infection, systemic corticosteroid requirement, drug/alcohol abuse) or laboratory abnormalities.
* Inability to wash-off specific medications (ask PI)
* Known hypersensitivity to cyclobenzaprine
* Others: seizure disorders, sleep apnea, continuous positive airway pressure (CPAP) use, BMI>40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Schmal, Study Director — Premier Research; Daniel J. Clauw, MD, Study Chair — Ann Arbor, MI
Locations (17):
- United States (17):
  - 107 Scripps Drive, Sacramento, California
  - Radiant Research, Inc., Denver, Colorado
  - 16176 Cortez Boulevard, Brooksville, Florida
  - 100 West Gore Street, Orlando, Florida
  - 3401 North Central Avenue, Chicago, Illinois
  - 71 Thomas Johnson Drive, Frederick, Maryland
  - 370 Faunce Corner Road, North Dartmouth, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - CRC of Jackson, LLC, Jackson, Mississippi
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - 1275 Olentangy River Road, Columbus, Ohio
  - 18660 Bagley Road, Middleburg Heights, Ohio
  - 1001 South Market Street, Mechanicsburg, Pennsylvania
  - 322 Memorial Drive, Greer, South Carolina
  - 1002 E. South Temple, Salt Lake City, Utah
  - 1951 152nd Place NE, Bellevue, Washington
  - 601 Broadway, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 205 patients were randomized to either TNX-102 SL or placebo; however, one patient was randomized in error (to the placebo group) and was not dispensed any study drug. Therefore, all disposition and safety tables are based on the safety population of 204 patients. Of these, 174 patients completed the study.
Pre-assignment Details: Screening for eligibility and washout of restricted medications.
Groups:
- TNX-102 SL 2.8 mg: 1 tablet of TNX-102 SL sublingually each day at bedtime for 12 weeks
- Placebo: 1 tablet of placebo sublingually each day at bedtime for 12 weeks.
Period: Overall Study
Arm/Group | TNX-102 SL 2.8 mg | Placebo
Started | 103 | 102
Completed | 89 | 85
Not Completed | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- TNX-102 SL 2.8 mg Tablets: 1 x TNX-102 SL 2.8mg Tablet taken sublingually each day at bedtime for 12 weeks.
  TNX-102 SL 2.8mg Tablets: Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
- Placebo: 1 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Placebo: Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks. (One patient randomized in error never received study drug and therefore is not included in this table.)
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo | Total
Number analyzed (Participants) | 103 | 101 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 96 | 199
  >=65 years | 0 | 5 | 5
Age, Continuous [Mean (Full Range); unit: years] | 50.7 [20 to 64] | 49.7 [19 to 65] | 50.2 [19 to 65]
Gender [Count of Participants; unit: Participants]
  Female | 96 | 98 | 194
  Male | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Weekly Average of Daily Pain Scores at Week 12
Description: Daily pain scores were assessed using a 24-hour recall response provided by each patient via an interactive voice response system (IVRS) daily telephone diary. Average daily pain was measured using an 11-point (0-10) numerical rating scale (NRS), with higher scores representing worse pain. Jump to control was used to replace missing data in each treatment arm.
Time Frame: Baseline, Week 12
Population: Patients in the Intention-to-treat (ITT) population: all randomized patients
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: 1 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Placebo: Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks.
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Number analyzed (Participants) | 103 | 102
units on a scale | -1.39 (0.253) | -0.95 (0.271)

2. Secondary Outcome: 30% Responder Analysis of IVRS NRS Pain Assessments at Week 12
Description: The weekly averages of daily pain scores were calculated using the daily, 24-hour-recall, IVRS NRS pain assessments.
  Patients who had at least a 30% improvement from baseline to week 12 in weekly average of daily pain scores were considered responders.
Time Frame: Baseline, Week 12
Population: Patients in the Intention-to-treat (ITT) population: all randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Number analyzed (Participants) | 103 | 102
percentage of participants | 34 | 20.6

3. Secondary Outcome: Change From Baseline to Week 12 in PROMIS T-score for Sleep Disturbance
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) sleep disturbance instrument consists of 8 items in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores are first synchronized prior to calculation of the total raw score. PROMIS scores are presented as T-scores in which the raw score has been rescaled into a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores represent more of the concept being measured (in this case, sleep disturbance).
Time Frame: Baseline, Week 12
Population: Patients in the Intention-to-treat (ITT) population: all randomized patients
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Number analyzed (Participants) | 103 | 102
units on a scale | -8.96 (0.993) | -5.13 (1.029)

4. Secondary Outcome: Patient Global Impression of Change (PGIC) Responder Status ("Very Much Improved" or "Much Improved" vs All Other Categories) at Week 12
Description: The PGIC is a 7-point scale (1=very much improved; 7=very much worse) that assesses the patient's perception of the overall change in his/her fibromyalgia symptoms since entering the study. Scores of 1 and 2 were considered responders.
Time Frame: Week 12
Population: Patients in the Intention-to-treat (ITT) population: all randomized patients
Measure: Number; unit: percentage of participants
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Number analyzed (Participants) | 103 | 102
percentage of participants | 30.1 | 16.7

5. Secondary Outcome: Change From Baseline to Week 12 in FIQ-R Total Score
Description: The Fibromyalgia Impact Questionnaire (revised) FIQ-R is made up of 3 domains: functional (9 questions), overall (2 questions) and symptoms (10 questions). All questions are based on an 11-point numerical rating scale (NRS) of 0-10, with 10 being "worst." Total FIQ-R scores can range from 0-100, with higher scores reflecting worsening status. The patient's total score on the FIQ-R was assessed at Visits 2, 3, 4, 5, and 6 (Week 12). Jump to control was used to replace missing data in each treatment arm.
Time Frame: Baseline, Week 12
Population: Patients in the Intention-to-treat (ITT) population: all randomized patients
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Number analyzed (Participants) | 103 | 102
units on a scale | -15.59 (2.079) | -8.54 (2.133)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: One placebo patient was never assigned study drug, thereby reducing the placebo group for safety analyses to 101 patients.
Arm/Group | TNX-102 SL 2.8 mg Tablets | Placebo
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/101
Other Adverse Events (participants affected / at risk) | 65/103 | 14/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNX-102 SL 2.8 mg Tablets (N=103) | Placebo (N=101)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL 2.8 mg Tablets (N=103) | Placebo (N=101)
hypoaesthesia oral (Gastrointestinal disorders) | 45 | 2
Nausea (Gastrointestinal disorders) | 5 | 2
Somnolence (Nervous system disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Product taste abnormal (General disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA in place with all study investigators.